CLINICAL TRIAL: NCT07196527
Title: Evaluation of the Clinical Efficacy of PURESSENTIEL Allergy Protection Nasal Spray (SNPA®) in House Dust Mite Allergic Rhinitis- ACARAY Study
Acronym: ACARAY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Puressentiel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CPP lDF 6 : 24.05823.000403
Record Dates: First submitted 2025-09-10; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Allergic Disorder of Respiratory System
Keywords: Allergic Rhinitis; Dust mite; Nasal Challenge
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: Patients will undergo a nasal mite challenge test, preceeded by the administration of either SPNA or placebo (saline solution)( D0). 15 days after the first test, they will perform a second test with the spray that was not administered on D0. Before, during and up to 4 hours after each nasal challenge test, the value of nasal inspiratory peak flow and a rhinitis score will be collected.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Puressentiel Protection Allergies nasal spray (SNPA) (Active Comparator): Each patient will receive two sprays per nostril of SPNA . Thirty minutes after administration of the sprays, a nasal provocation test with Dermatophagoides pteronyssinus (LETI Pharma) will be performed according to the recommendations of the European Academy of Allergy and Clinical Immunology (EAACI).
  For the nasal provocation test, the patient will be seated and at rest for 10 minutes before the start of the test. The patient will be in apnea, with their mouth open. A spray of 0.3 HEP/ml will be administered into each nostril.
  Interventions: Device: Puressentiel Allergy Protection Nasal Spray
- Saline spray (Placebo Comparator): Placebo Comparator: Saline spray Arm Description: Each patient will receive two sprays per nostril of placebo (saline solution). Thirty minutes after administration of the sprays, a nasal provocation test with Dermatophagoides pteronyssinus (LETI Pharma) will be performed according to the recommendations of the European Academy of Allergy and Clinical Immunology (EAACI). For the nasal provocation test, the patient will be seated and at rest for 10 minutes before the start of the test. The patient will be in apnea, with their mouth open. A spray of 0.3 HEP/ml will be administered into each nostril.
  Interventions: Device: Saline spray (0.65%)

INTERVENTIONS:
Device: Puressentiel Allergy Protection Nasal Spray — Crossover study after nasal provocation test (Dermatophagoides pteronyssinus)
  Arms: Puressentiel Protection Allergies nasal spray (SNPA)
Device: Saline spray (0.65%) — Crossover study after nasal provocation test (Dermatophagoides pteronyssinus)
  Arms: Saline spray

SUMMARY:
Justification of the relevance of the research:

Patients suffering from allergic rhinitis are looking for several therapeutic options to control their symptoms. Although etiological treatment is based on allergen immunotherapy, and most prescribed symptomatic therapies include antihistamines and/or topical corticoids, patients tend to self-medicate and seek different options, also choosing non-pharmacological approaches, particularly when symptoms are milder; nevertheless, accurate and reliable information on non-conventional therapies remains limited.

Main research hypothesis and objectives:

The present study, will prospectively investigate the potential role of Puressentiel® Protection Allergies nasal spray (SNPA) in patients suffering from house dust mite allergic rhinitis.

Assessment of the benefits and risks of the research, including the expected benefits for the people who undergo the research and the foreseeable risks associated with the research treatment and investigative procedures:

No individual benefit is expected. With regard to possible indirect benefits, this study could help to propose a natural, alternative solution to symptomatic medication for the symptoms of allergic rhinitis in mite-allergic patients. The main risks of this study are those linked to the performance of the nasal challenge test, i.e. the appearance of symptoms of allergic rhinitis.

Justification for the inclusion of persons covered by articles L.1121-5 to L.1121-8 and L.1122-1-2 of the French Public Health Code (e.g. minors, protected adults, etc.) and procedure implemented to inform and obtain the consent of these persons or their legal representatives.

Subjects over 18 years of age will be included in this project. People under court protection, guardianship or curatorship are excluded from this research.

Description of the recruitment process:

Patients are recruited at the time of consultation in the Division of Allergology, Department of Pneumology, Allergology and Thoracic Oncology, Hôpital Arnaud de Villeneuve - CHU de Montpellier, whatever the reason for the consultation (respiratory allergies, food allergies, drug allergies, skin allergies). Patients will be given a period of reflection before confirming their participation by signing an express consent form.

Investigation procedures carried out:

After a rhinitis and possibly asthma control test, patients will undergo a nasal mite challenge test, preceeded by the administration of either SPNA or placebo (saline solution)( D0). 15 days after the first test, a second test will be performed with the spray that was not administered on D0. Before, during and up to 4 hours after each nasal challenge test, the value of nasal inspiratory peak flow and a rhinitis score will be collected.

Justification of whether or not there is: (1) a prohibition on simultaneous participation in other research; (2) an exclusion period during which participation in other research is prohibited/ Given the need to stop anti-allergy treatments before and during the study; participation in another study is not permitted 7 days before the start of the present study and 7 days after its end (exclusion period).

Terms and amount of compensation for research participants Researchers will be compensated up to €500. Anticipated number of people to be included in the research 20 (twenty)

DETAILED DESCRIPTION:
Main objective:

Testing the protective effect of SNPA on the nasal inflammatory allergic response in subjects with allergic rhinitis caused by dust mites.

The main objective of this clinical investigation is to evaluate the reduction in rhinoconjunctivitis symptoms following a nasal provocation test (Dermatophagoides pteronyssinus) performed after administration of Puressentiel Allergy Protection Nasal Spray, compared to those developed after administration of a placebo.

Secondary objectives

* Evaluate the difference in terms of nasal obstruction, measured by inspiratory nasal peak flow (INPF), after administration of the protective nasal spray and after placebo.
* Evaluate the duration of symptoms after performing the TPN and check whether there is a difference after the tests performed with the SPNA and with the placebo.

Méthodology

* 1 Type of study This is a prospective, single-center, crossover, randomized, double-blind, placebo-controlled study in adult subjects with allergic rhinitis caused by dust mites.
* 2 Main evaluation criteria The primary endpoint will be the difference between the validated symptom score for nasal provocation tests after performing the test with SPNA and with placebo.
* 3 Secondary evaluation criteria

  * Difference between the value obtained with PFIN before TPN and after TPN and the difference between the results obtained when SPNA and placebo were administered beforehand.
  * Difference between the duration of symptoms appearing after TPN with SPNA and with placebo
* 4 Scheduled visits and examinations

Two visits are planned, with at least 15 days (+7) between visits (washout period). During each of the two visits, patients will undergo a clinical assessment and nasal provocation tests. Before the tests begin, the clinical assessment will include:

* Rhinitis control test (ARCT) and asthma control test (ACT), if applicable;
* Nasal and conjunctival symptom score ;
* Nasal inspiratory peak flow (NIPF).

Each patient will receive two sprays per nostril of SPNA or placebo (saline solution), depending on randomization. Those who received SPNA during the visit on Day 0 will receive the placebo on Day 15, and vice versa. Thirty minutes after the administration of the spray, a nasal provocation test with Dermatophagoides pteronyssinus (LETI Pharma) will be performed according to the recommendations of the European Academy of Allergy and Clinical Immunology (EAACI).

For the nasal provocation test, the patient will be seated and at rest for 10 minutes before the start of the test. They will be informed about the test procedure, with particular emphasis on the fact that they must not breathe through their nose or sniff during the administration of the solutions. They will be warned of the various symptoms that may occur: tingling, sneezing, nasal discharge, and nasal congestion. The patient will be in apnea, with their mouth open. A spray of 0.3 HEP/ml will be administered into each nostril, followed by the placement of a nose clip, which will be removed after 10 minutes. A second dose of 3 HEP/ml will then be administered, following the same procedure as before. After 10 minutes, the nose clip will be removed. New assessments of nasal symptom scores and PFIN will be performed between the two doses of TPN, at the end of TPN, and 30, 60, 120, and 240 minutes after TPN.

ELIGIBILITY:
Inclusion Criteria:General inclusion criteria:

* The patient must have given their express consent to participate in the study.
* The patient must be affiliated with or a beneficiary of a health insurance plan.
* The patient is at least 18 years of age.

Inclusion criteria for the target population:

* Patients who have already consulted the allergy department at Montpellier University Hospital.
* Patients suffering from perennial rhinitis (or rhino-conjunctivitis) caused by dust mites, diagnosed more than one year ago.
* In the case of asthmatic patients, asthma must be under control.
* Patients who have been able to stop all treatment with antihistamines or nasal corticosteroids for one week prior to the start of the study (7 days and 1 month, respectively).
* Patients covered by social security.

Exclusion Criteria:5.4 Exclusion Criteria

General exclusion criteria:

* The patient is in a period of exclusion determined by a previous study.
* The patient is under judicial protection, guardianship, or curatorship.
* The patient is a minor.
* The patient is not fluent in French.

Exclusion criteria regarding interfering diseases or conditions:

* The patient is pregnant and/or breastfeeding.
* Patient sensitized to a perennial allergen in addition to dust mites.
* Patient sensitized to a seasonal allergen, during the allergen's peak pollen season.
* Patient who has had a viral infection within 4 weeks prior to the provocation test.
* Patient treated or undergoing treatment with allergen immunotherapy.
* Patient treated with antihistamines (7-day washout period) or nasal corticosteroids (1-month washout period).
* Patients with severe uncontrolled asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Allergic Rhinitis Control Test (ARCT) | ARCT will be recorded 30, 60, 120 and 240 minutes after the nasal provocation test
  A nasal provocation test with Dermatophagoides pteronyssinus (LETI Pharma) will be performed according to the recommendations of the European Academy of Allergy and Clinical Immunology (EAACI) after which ARCT will be recorded;

SECONDARY OUTCOMES:
Nasal and conjunctival symptom score | Nasal and conjunctival symptom score will be recorded 30, 60, 120 and 240 min after the nasnal provocative test
Nasal Inspiratory Peak Flow | Nasal Inspiratory Peak Flow will be recorded, 30, 60, 120 and 240 min after the nasal provocative test

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Demoly, MD,PhD, Principal Investigator — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: Undecided